CLINICAL TRIAL: NCT07040735
Title: The Effect of Low-Flow Anesthesia on Hemodynamics in Open-Heart Surgery
Brief Title: Low-Flow Anesthesia and Open-Heart Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Çağrı Özdemir (Other)
Responsible Party: Sponsor-Investigator, Çağrı Özdemir, asst. prof., Gazi University
Organization: Gazi University (Other)
Other Study IDs: 2025-146
Record Dates: First submitted 2025-06-06; First posted 2025-06-27 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Low-flow Anesthesia; Hemodynamics; Open-heart Surgery
Keywords: Low-flow anesthesia; Hemodynamics; Open-heart surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Followed using Bispectral Index (BIS) with 4% Sevoflurane and fresh gas flow set at 0.5 L/min
- Group 2: Followed using Minimum Alveolar Concentration (MAC) with 4% Sevoflurane and fresh gas flow set at 0.5 L/min
- Group 3: Followed using BIS with 4% Sevoflurane and fresh gas flow set at 1 L/min
- Group 4: Followed using MAC with 4% Sevoflurane and fresh gas flow set at 1 L/min

SUMMARY:
Low-flow anesthesia (LFA) is a technique in which at least 50% of the exhaled air, after carbon dioxide absorption, is mixed with a certain amount of fresh gas and returned to the patient during the next inspiration. In 1974, R. Virtue defined minimal flow anesthesia (MFA) as 0.5 L/min. In 1984, Baker and Simionescu classified LFA as 0.5-1 L/min and MFA as 0.25-0.5 L/min. The aim of this study is to investigate whether there are hemodynamic differences between open-heart surgery cases performed with LFA at different fresh gas flow rates.

ELIGIBILITY:
Inclusion Criteria:

-≥18 years and scheduled for open-heart surgery patients

-ASA I-II-III-IV physical class

Exclusion Criteria:

* Emergency cases
* Patients under 18 years of age
* Patients who have had open heart surgery before
* Patients for whom the use of inhaled anesthetic agents is contraindicated
* Patients who do not sign a voluntary consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ≥18 years and scheduled for open-heart surgery patients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
physiological parameter ; heart rate | Intraoperatively
  Heart rate will be recorded every 10 minutes, expressed as beats per minute, starting before induction and including the sternotomy and pericardiotomy periods.
physiological parameter; systolic/diastolic blood pressure | Intraoperatively
  Systolic and diastolic blood pressure will be recorded every 10 minutes in mmHg, starting before induction and including the sternotomy and pericardiotomy periods.
physiological parameter; SpO2 | Intraoperatively
  SpO2 will be recorded as a percentage every 10 minutes, starting before induction and including the sternotomy and pericardiotomy periods.
Monitoring parameter; Bispectral Index (BIS) | Intraoperatively
  The BIS value will be recorded numerically every 10 minutes, starting from before induction and including the sternotomy and pericardiotomy periods.
Monitoring parameter; Minimum alveolar concentration (MAC) | Intraoperatively
  The MAC value will be recorded numerically every 10 minutes, starting from before induction and including the sternotomy and pericardiotomy periods.

SECONDARY OUTCOMES:
Preoperative data; ASA classification | 24 hours before surgery
  During the preoperative period, the patient's ASA classification will be recorded as I, II, III, IV.
Preoperative data | 24 hours before surgery
  In the preoperative period, the degree of valve dysfunction (such as I.degree TY, II.degree MY) of the patients will be recorded.
Preoperaitive data | 24 hours before surgery
  In the preoperative period, the patient's ejection fraction will be recorded as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No